CLINICAL TRIAL: NCT05028114
Title: A Phase 1, Three-part, Part-randomised, Study to Evaluate the Pharmacokinetics, Safety, and Tolerability of Different Formulations of Tricaprilin, to Include Single-dose, Food Effect, and Titration Tolerability, in Healthy Participants
Brief Title: Tricaprilin Liquid Formulation PK Study
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Part 1 was completed, Part 2 and Part 3 of the study were not conducted under this study protocol due to subject recruitment difficulty.
Sponsor: Cerecin (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: AC-21-025
Record Dates: First submitted 2021-08-19; First posted 2021-08-31 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-10

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — AC-1202

STUDY DESIGN:
Intervention Model Description: This is a three-part study.
  Part 1 (Formulation Optimisation): Participants will be assigned to all 4 different formulations of tricaprilin, with randomization to one of 4 sequences with a 2-day washout in between different formulations. There are 2 series in this part.
  Part 1 (Food Effect): Participants will be administered to 1 formulation of tricaprilin. There are 2 series in this part.
  Part 2 (Placebo Assessment): Participants will be randomised to 1 of 2 sequences (tricaprilin formulation - matching placebo; matching placebo - tricaprilin formulation) with a 2-day washout between periods.
  Part 3 (Titration Tolerability): Participants will be administered to either tricaprilin or a matching placebo.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Part 1 (Formulation Optimisation) (Experimental): Study drug administered orally after an overnight fast (minimum 8 hours). A standard breakfast will be provided 30 minutes after study drug administration. There will be 4 different formulations of the study drug and participants will be randomised to one of 4 sequences. There will be a washout of 2 days between each administration.
  Interventions: Drug: AC-1202; Drug: AC-OLE-01; Drug: AC-OLE-02; Drug: AC-OLE-03; Drug: AC-OLE-04; Drug: AC-OLE-05; Drug: AC-OLE-06; Drug: AC-OLE-07; Drug: AC-OLE-08; Drug: AC-OLE-09; Drug: AC-OLE-010
- Part 2 (Placebo Assessment) (Experimental): Study drug administered orally after an overnight fast (minimum 8 hours). A standard breakfast will be provided either 30 minutes before or after study drug administration, depending on the results of the food effect assessment.
  Participants are randomised to 1 of 2 sequences (tricaprilin formulation - matching placebo; matching placebo - tricaprilin formulation) with a 2-day washout between periods.
  Interventions: Drug: AC-OLE-P
- Part 3 (Titration Tolerability) (Experimental): Study drug administered orally after an overnight fast (minimum 8 hours). A standard breakfast will be provided either 30 minutes before or after study drug administration, depending on the results of the food effect assessment.
  Participants will be randomised to either study drug or the matching placebo.
  Interventions: Drug: AC-OLE-P

INTERVENTIONS:
Drug: AC-1202 — Tricaprilin formulated as AC-1202
  Arms: Part 1 (Formulation Optimisation)
Drug: AC-OLE-01 — Tricaprilin Formulation
  Arms: Part 1 (Formulation Optimisation)
Drug: AC-OLE-02 — Tricaprilin Formulation
  Arms: Part 1 (Formulation Optimisation)
Drug: AC-OLE-03 — Tricaprilin Formulation
  Arms: Part 1 (Formulation Optimisation)
Drug: AC-OLE-04 — Tricaprilin Formulation
  Arms: Part 1 (Formulation Optimisation)
Drug: AC-OLE-05 — Tricaprilin Formulation
  Arms: Part 1 (Formulation Optimisation)
Drug: AC-OLE-06 — Tricaprilin Formulation
  Arms: Part 1 (Formulation Optimisation)
Drug: AC-OLE-07 — Tricaprilin Formulation
  Arms: Part 1 (Formulation Optimisation)
Drug: AC-OLE-08 — Tricaprilin Formulation
  Arms: Part 1 (Formulation Optimisation)
Drug: AC-OLE-09 — Tricaprilin Formulation
  Arms: Part 1 (Formulation Optimisation)
Drug: AC-OLE-010 — Tricaprilin Formulation
  Arms: Part 1 (Formulation Optimisation)
Drug: AC-OLE-P — Placebo to tricaprilin formulation
  Arms: Part 2 (Placebo Assessment); Part 3 (Titration Tolerability)

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetics, safety, and tolerability of new liquid formulations of tricaprilin, with the aim of finding a suitable formulation to advance in development. This is a three-part, part-randomised study that include single-dose, food effect, and titration tolerability in up to 80 healthy participants.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be 18 to 65 years of age inclusive, at the time of signing the informed consent.
* Participants who are overtly healthy (in the opinion of the Investigator) as determined by medical evaluation including medical history, physical examination, laboratory tests, and cardiac monitoring
* Body weight ≥45 kg and body mass index (BMI) within the range 18.0 - 32.0 kg/m2 (inclusive).
* Male and female
* Agrees to comply with study procedures including blood draws, confinement to clinic, meal requirements
* Continuous non-smoker or infrequent smoker (no more than 10 cigarettes per week for at least 3 months prior to Screening)

Exclusion Criteria:

* History of, or current gastrointestinal (GI) conditions constituting a risk when taking the study treatment; or interfering with the interpretation of data, based on the Investigator's judgement
* Past or intended use of over-the-counter or prescription medication including herbal medications within 7 days prior to dosing (paracetamol/acetaminophen [up to 2 g per day], hormone replacement therapy and hormonal contraception are permitted).
* Participants on a ketogenic diet, low-fat diet or actively using medium chain triglycerides, ketone esters, or other ketogenic products.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2021-08-31 (Actual); Primary Completion 2022-03-18 (Actual); Study Completion 2022-07-19 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve (AUC) of total ketones (β-hydroxybutyrate and acetoacetate) after single-dose administration of tricaprilin and placebo formulations (Part 1, Part 2) | 0 to 8 hours post-dose
  AUC will be calculated from PK concentrations of total ketones (B-hydroxybutyrate and Acetoacetate)
Maximum observed concentration (Cmax) of total ketones (β-hydroxybutyrate and acetoacetate) after single-dose administration of tricaprilin and placebo formulations (Part 1, Part 2) | 0 to 8 hours post-dose
  Cmax will be calculated from PK concentrations of total ketones (B-hydroxybutyrate and Acetoacetate)
Time of maximum concentration (Tmax) of total ketones (β-hydroxybutyrate and acetoacetate) after single-dose administration of tricaprilin and placebo formulations (Part 1, Part 2) | 0 to 8 hours post-dose
  Tmax will be calculated from PK concentrations of total ketones (B-hydroxybutyrate and Acetoacetate)

SECONDARY OUTCOMES:
Incidence of treatment emergent adverse events | Baseline to end of treatment period
  Adverse event incidence will be tabulated
Gastrointestinal side effects of single-dose administration of each of tricaprilin formulations and the placebo formulation (Parts 1, 2) assessed using the Baxter Retching Faces Scale | Pre-dose, 0.5, 1, 1.5, 2, 3 hours post-dose
  The Baxter Retching Faces Scale is a pictorial scale rated from 0 to 10, with 6 faces depicting level of nausea/gastrointestinal discomfort.
Gastrointestinal side effects of single-dose administration of each of tricaprilin formulations and the placebo formulation (Parts 1, 2) assessed using the Pain Numerical Rating Scale | Pre-dose, 0.5, 1, 1.5, 2, 3 hours post-dose
  The Pain Numerical Rating Scale 10-point numeric rating scale with participants instructed to rate any abdominal pain from 0 (no pain) to 10 (worst possible pain)
Area under the concentration-time curve (AUC) of total ketones (β-hydroxybutyrate and acetoacetate) of tricaprilin and placebo formulations following a titration scheme (Part 3) | Days 15 and 21: 0 to 8 hours post-dose; Day 27: 0 to 24 hours post-dose
  AUC will be calculated from PK concentrations of total ketones (B-hydroxybutyrate and Acetoacetate)
Maximum observed concentration (Cmax) of total ketones (β-hydroxybutyrate and acetoacetate) of tricaprilin and placebo formulations following a titration scheme (Part 3) | Days 15 and 21: 0 to 8 hours post-dose; Day 27: 0 to 24 hours post-dose
  Cmax will be calculated from PK concentrations of total ketones (B-hydroxybutyrate and Acetoacetate)
Time of maximum concentration (Tmax) of total ketones (β-hydroxybutyrate and acetoacetate) of tricaprilin and placebo formulations following a titration scheme (Part 3) | Days 15 and 21: 0 to 8 hours post-dose; Day 27: 0 to 24 hours post-dose
  Tmax will be calculated from PK concentrations of total ketones (B-hydroxybutyrate and Acetoacetate)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Cerecin
Locations (1):
- CMAX, Adelaide, South Australia, Australia

IPD SHARING:
Plan to Share IPD: No